CLINICAL TRIAL: NCT01707589
Title: Noninvasive Monitoring of Vital Signs in Neonates
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pediatric Elfi-Monitor
Record Dates: First submitted 2012-09-10; First posted 2012-10-16 (Estimated); Last update posted 2013-02-12 (Estimated); Status verified 2013-02

CONDITIONS: Admission to the NICU and Need for Physiological Monitoring.
Keywords: monitoring; heart rate; respiration rate; temperature; motion; noninvasive; physiologic parameters; NICU

ARMS (1):
- Neonates admitted to the NICU (Experimental): Neonates admitted to the NICU for a variety of medical reasons will be the cohort group. Those whose parents give informed consent will compose the subjects of the study
  Interventions: Device: The new sensor is not on the market. We have named it Elfi-sensor.

INTERVENTIONS:
Device: The new sensor is not on the market. We have named it Elfi-sensor. — Participating subjects will be monitored for one hour with a noninvasive sensor.The noninvasive sensor, the size of a penny, will be affixed to the skin, above the umbilicus, with pediatric adhesive tape. The monitor will record continuously the heart rate, cardiac rhythm, respiratory rate and body motion.

SUMMARY:
the investigators are assessing a non-invasive monitor based on dynamic light scattering that measures pulse rate and respiration rate. The monitor also will be equipped with a temperature sensor and a motion sensor. This monitor will allow multi-parametric measurements in neonates in a simple and noninvasive manner.

DETAILED DESCRIPTION:
Monitoring vital signs in neonates is important. This currently is done with multiple standard clinical monitors. the investigators are developing a very small (coin-sized) sensor that can measure pulse rate, respiratory rate, temperature and body motion. the investigators propose to test our sensor against standard monitoring techniques in neonates in a neonatal ICU (NICU).

The monitor, called ELFI-monitor, is based on dynamic light scattering. A low-power laser beams light into the skin, and the red blood cells in the underlying skin return the light which is recorded in a light sensor. The movement of the red blood cells is affected by the rhythmic cardiac contractility. in this manner, heart rate and rhythm can be assessed. The ELFI monitor also contains an embedded temperature probe and a miniature 3-D motion sensor, allowing capture of additional parameters.

Methods:

the investigators plan to study 100 neonates admitted to the NICU of Meir Hospital Center. These infants are routinely monitored with standard equipment including ECG, oximeter, temperature, and respiratory monitors. the investigators will simultaneously monitor these children with the ELFI monitor, recording pulse rate, cardiac rhythm, respiratory rate, skin temperature and body motion. Recordings will be conducted for a one-hour period on each subject. Data recordings from the ELFI sensor will be compared to the readouts of the conventional monitors used on the patient. It is important to emphasize that the data recordings of the ELFI sensor will not affect clinical decisions in any manner, but will merely be recorded for comparison with conventional sensors.

ELIGIBILITY:
Inclusion Criteria:

* All neonates admitted the Meir Hospital center NICU
* Parents provide informed consent

Exclusion Criteria:

* Neonates with skin disease

Ages: 1 Day to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2013-05; Primary Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Comparison of data collected from ELFI sensor to standard monitors | 6 months
  the investigators are comparing the data recoded by the new sensor to that recorded by conventional sensors during a period of one hour in the NICU. The data recorded by the new sensor will not be used for clinical decision making.

CONTACTS AND LOCATIONS:
Overall Officials: Sofia Bauer-rosek, MD, Principal Investigator — Meir Medical Center
Locations (1):
- Neonatal department Meir Medical Center, Kfar Saba, Israel